CLINICAL TRIAL: NCT01020266
Title: Clinical Trial of Cerebral Protective Effects of Repeated Electroacupuncture Pretreatment in Heart Valve Replacement Surgery
Brief Title: Neuroprotective Study of Electroacupuncture Pretreatment in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJMZK015
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2009-11

CONDITIONS: Stroke; Brain Injuries
Keywords: brain protection; cardiac surgery; heart valve replacement; electroacupuncture; pretreatment; preconditioning; Thoracic Surgery
MeSH Terms: conditions — Stroke; Brain Injuries | interventions — Acupuncture Therapy; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture (Active Comparator)
  Interventions: Procedure: Electroacupuncture pretreatment
- Control (Sham Comparator)
  Interventions: Procedure: non electroacupuncture stimulation

INTERVENTIONS:
Procedure: non electroacupuncture stimulation — The same procedure as electroacupuncture except stimulation
  Arms: Control
Procedure: Electroacupuncture pretreatment — According to the theory of traditional Chinese medicine, Baihui(GV20) acupoint was chosen and the acupuncture points were identified according to traditional anatomical localization. Once insertion was made at the acupuncture point, the needle was stimulated electrically with the intensity of 0.8-1.9 mA and frequency of 5/30 Hz for 30 min per day using an Electronic Acupuncture Treatment Instrument for 5 consecutive days before the heart valve replacement surgery．
  Other Names: Acupuncture; preconditioning; electric stimulation
  Arms: Electroacupuncture

SUMMARY:
The purpose of this study is to evaluate the neuroprotective effect of electroacupuncture pretreatment in patients undergoing cardiac surgery as an preventive sequela in a randomized and controlled clinical trial. In addition, to investigate the role of inflammatory responses in the precess of the protection.

DETAILED DESCRIPTION:
Heart valve replacement surgery has been proved to be an effective method in treating both regenerative and rheumatic valve disease. Current studies showed that cardiopulmonary bypass (CPB) and operation related cerebral injury is associated with worse patient morbidity and mortality after elective valve replacement surgery. Recently, Electroacupuncture (EA) pretreatment was proved to produced cerebral protective effects by mimicking ischemic preconditioning in animal models. However, the evidence that EA pretreatment can improve the clinical outcomes such as mortality and morbidity, is still lacking. The investigators perform a randomized controlled study to evaluate that EA pretreatment can improve the outcomes of cardiac surgery.

Purpose:

The purpose of this study is to examine if EA pretreatment can decrease the mortality and postoperative cerebrovascular complications in patients undergoing cardiac surgery. The effect will be assessed by mortality, scores of neurological defect, post operative cognitive dysfunction and stroke.

Methods:

Study patients will be randomized to cardiac surgery with EA pretreatment or conventional cardiac surgery in the Department of cardiovascular surgery, Xijing Hospital. EA pretreatment is performed at Baihui acupoint 30 min per day 5 consecutive days before the heart valve replacement surgery．Primary study outcome is cerebrovascular complications within 6 postoperative months. Secondary outcomes include the S-100B and NSE blood level measured during the first 72 hours of surgery follow-up, the several cytokines, including TNF-a, IL-8, IL-6, IL-10 and HMGB-1 blood level measured during the first 7 days of surgery follow-up, all cardiovascular haemodynamic parameters as measured by a pulmonary artery catheter, the length of intensive care unit (ICU) stay and length of postoperative hospital stay.

ELIGIBILITY:
This study enrolls a group of 40-65years patients who have heart valve disease who need valve replacement.

Inclusion Criteria:

* patients who have the indication for aortic or mitral valve replacement
* patients would like to accept the follow-up and sign the informed consent
* patients with heart function of NYHA I-III degree.

Exclusion Criteria:

* pregnant or nursing women
* comorbid with coronary artery disease
* patients with heart function of NYHA IV degree
* renal dysfunction with serum creatinine level>or=2mg/dl(177umol/L)
* anticipated life span < 12 months
* enrollment in other clinical trials at the same time not reaching the primary endpoint and probably interference the present trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular complications and Score of neurological defect | before treatment, after the first treatment, 7, 28days after treatment and follow up at 6 months after treatment

SECONDARY OUTCOMES:
The S-100B and NSE blood level | before treatment, after the last treatment, before surgery, and the first 72 hours of surgery follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Aideng Weng, Ph.D., Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China